CLINICAL TRIAL: NCT01822067
Title: Effects of Maternal Body Composition on Offspring Brain Structure and Function
Status: Active, not recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 134776
Record Dates: First submitted 2013-02-26; First posted 2013-04-02 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Brain Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weight- Non Maternal obesity: Full-term neonates at 2 weeks of age born to normal weight mothers
- Obese- Obese Mothers: Full-term neonates at two weeks of age born of obese mothers

SUMMARY:
The specific aim of this study is to use MRI methods to evaluate and compare brain structure and function in two groups of full-term neonates at two-weeks of age: those born of obese mothers and those born to normal weight mothers.

ELIGIBILITY:
Inclusion Criteria:

* the participant must be enrolled in the Arkansas Children's Nutrition Center (ACNC) Glowing study and be about 2 weeks of age +/- 3days

Exclusion Criteria:

* none specified

Ages: 11 Days to 17 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full term neonates born from obese or lean mothers enrolled in the Glowing study (IRB#110889)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Brain Structure | Age 2 weeks
  We will use high resolution volumetric magnetic resonance imaging (MRI) and Diffusion tensor imaging (DTI) to measure the brain structure of 2 week old infants

SECONDARY OUTCOMES:
Brain Function | Age 2 weeks
  We will use high resolution Resting state functional magnetic resonance imaging (rsfMRI) to measure the brain function of 2 week old infants

CONTACTS AND LOCATIONS:
Overall Officials: Xiawei Ou, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States